CLINICAL TRIAL: NCT02419326
Title: Uniting Couples In the Treatment of Eating Disorders (UNITE): Pilot Study for a Couple-based Intervention for Binge-eating Disorder
Brief Title: Uniting Couples In the Treatment of Eating Disorders (UNITE)
Acronym: UNITE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: The Hilda & Preston Davis Foundation (Other); Global Foundation for Eating Disorders (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14-1599
Record Dates: First submitted 2015-03-31; First posted 2015-04-17 (Estimated); Last update posted 2016-10-27 (Estimated); Status verified 2016-10

CONDITIONS: Binge-eating Disorder; Eating Disorder
Keywords: couples; relationships; binge eating; eating disorder; couple therapy
MeSH Terms: conditions — Binge-Eating Disorder; Feeding and Eating Disorders; Bulimia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Couples (Experimental): The patient and their significant other receive psychotherapy treatment for the patient's BED.
  Interventions: Behavioral: Psychotherapy treatment

INTERVENTIONS:
Behavioral: Psychotherapy treatment — UNITE is a manualized, 22-session CBCT (cognitive behavioral couples therapy) intervention that engages the couple to target the core psychopathology of BED and address the uniquely challenging stress that BED places on intimate relationships.

SUMMARY:
The purpose of this study is to test the feasibility, acceptability, and preliminary efficacy of a novel couple-based intervention for binge-eating disorder (BED).

DETAILED DESCRIPTION:
Although current individual treatments exist for BED (e.g., cognitive-behavior therapy and interpersonal psychotherapy) about 20% of individuals who complete treatment and who are abstinent from binge eating post-treatment relapse within one year. In addition, dropout of BED treatment is high (approximately 10 - 33%), indicating that a significant number of individuals with BED fail to achieve relief from their symptoms. Couple-based interventions, which enlist the support of a partner into the treatment setting, are effective for treating anxiety and depression--frequently comorbid conditions with BED. Preliminary findings of couple-based treatment for anorexia nervosa suggests it assists in reducing drop out and improving outcome. Thus, the investigators developed a novel couple-based intervention for adult BED (UNITE-BED Edition) and plan to investigate it in an open treatment trial to examine it's feasibility, acceptability, and preliminary efficacy. Both patients and partners will be involved in all psychotherapy sessions of the treatment. Couples' progress will be followed for three months after completion of active treatment.

ELIGIBILITY:
Inclusion Criteria:

Participant with BED:

1. Subject currently meets criteria for BED or sub-threshold symptoms, according to the Diagnostic and Statistical Manual of Mental Disorders (5th Ed)
2. Concurrent outpatient therapy and medical monitoring
3. Health insurance coverage

Both members of the couple:

1. English speaking and able to read
2. Involved in a committed relationship for at least 6 months regardless of sexual orientation (couple is not required to live together)
3. Willing to participate in treatment

Exclusion Criteria:

Participant with BED:

1) Post-bariatric

Both members of the couple:

1. Alcohol or drug dependence in the last year
2. Current significant suicidal ideation
3. Severe depression that would seriously interfere with functional capacity
4. Developmental disability that would impair the ability to benefit from intervention
5. Any psychosis, schizophrenia, or bipolar I disorder, unless stably remitted on maintenance therapy for at least 1 year
6. Moderate to high levels of physical violence from either partner as reported on the Conflict Tactics Scale-2 at pre-treatment
7. Unwillingness to forgo non-protocol concurrent couples therapy
8. Previously participated in the preliminary couples treatment study UCAN: Uniting Couples (in the treatment of) Anorexia Nervosa (NCT01740752)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2014-09; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Total score at Post-treatment of the Client Satisfaction Questionnaire-8 (CSQ-8)- Patient | Post-treatment (on average 6 months after beginning treatment)
  8-item self-report scale assessing the effectiveness of, and satisfaction with, content and format of treatment.
Total score at Post-treatment of the Client Satisfaction Questionnaire-8 (CSQ-8)- Partner | Post-treatment (on average 6 months after beginning treatment)
  8-item self-report scale assessing the effectiveness of, and satisfaction with, content and format of treatment.

SECONDARY OUTCOMES:
Number of patients with binge-eating remission (0 objective binge episodes over last 28 days) at post-treatment determined by Eating Disorder Examination (EDE) | Post-treatment (on average 6 months after beginning treatment)
  Clinical interview used to establish the diagnosis of BED and eating disorder severity. It inquires about the number of objective and subjective binge episodes and days over the 28 days prior to the assessment period.
Number of patients with binge eating remission (0 objective binge-eating episodes in last 28 days) at 3-month follow-up determined by the Eating Disorder Examination (EDE) | 3-Month Follow-up
  Clinical interview used to establish the diagnosis of BED and eating disorder severity. It inquires about the number of objective and subjective binge episodes and days over the 28 days prior to the assessment period.
Change from Baseline to Post-Treatment in the Eating Disorder Examination (EDE) Binge Eating Episode Frequency Score- Patient | Baseline, Post-Treatment (on average 6 months after beginning treatment)
  Clinical interview used to establish the diagnosis of BED and eating disorder severity. It inquires about the number of objective and subjective binge episodes and days over the 28 days prior to the assessment period.
Change from Baseline to 3-Month Follow-up in the Eating Disorder Examination (EDE) Binge Eating Episode Frequency Score- Patient | Baseline, 3-Month Follow-up
  Clinical interview used to establish the diagnosis of BED and eating disorder severity. It inquires about the number of objective and subjective binge episodes and days over the 28 days prior to the assessment period.
Change from Baseline to Post-Treatment in the Eating Disorder Examination (EDE) Number of Days Binge Eating Score- Patient | Baseline, Post-Treatment (on average 6 months after beginning treatment)
  Clinical interview used to establish the diagnosis of BED and eating disorder severity. It inquires about the number of objective binge and subjective episodes and days over the 28 days prior to the assessment period.
Change from Baseline to 3-Month Follow-up in the Eating Disorder Examination (EDE) Number of Days Binge Eating Score- Patient | Baseline, 3-Month Follow-up
  Clinical interview used to establish the diagnosis of BED and eating disorder severity. It inquires about the number of objective and subjective binge episodes and days over the 28 days prior to the assessment period.
Change from Baseline to Post-Treatment in the Binge Eating Scale (BES) Binge Eating Symptom Severity- Patient | Baseline, Post-Treatment (on average 6 months after beginning treatment)
  16-item self-report scale assessing the presence of specific binge-eating behaviors commonly observed in individuals with BED.
Change from Baseline to 3-Month Follow-up in the Binge Eating Scale (BES) Binge Eating Symptom Severity- Patient | Baseline, 3-Month Follow-up
  16-item self-report scale assessing the presence of specific binge-eating behaviors commonly observed in individuals with BED.
Change from Baseline to Post-Treatment in the Yale-Brown Obsessive Compulsive Scale Modified for Binge Eating (YBOCS-BE) Total Score- Patient | Baseline, Post-Treatment (on average 6 months after beginning treatment)
  Clinical interview used to assess obsessiveness of binge-eating thoughts and compulsiveness of binge-eating behaviors.
Change from Baseline to 3-Month Follow-up in the Yale-Brown Obsessive Compulsive Scale Modified for Binge Eating (YBOCS-BE) Total Score- Patient | Baseline, 3-Month Follow-up
  Clinical interview used to assess obsessiveness of binge-eating thoughts and compulsiveness of binge-eating behaviors.
Change from Baseline to Post-Treatment in the Eating Disorder Examination (EDE) Total Score- Patient | Baseline, Post-Treatment (on average 6 months after beginning treatment)
  Clinical interview used to establish the diagnosis of BED and eating disorder severity. It inquires about eating disorder symptoms and severity over the 28 days prior to the assessment period.
Change from Baseline to 3-Month Follow-up in the Eating Disorder Examination (EDE) Total Score- Patient | Baseline, 3-Month Follow-up
  Clinical interview used to establish the diagnosis of BED and eating disorder severity. It inquires about eating disorder symptoms and severity over the 28 days prior to the assessment period.
Change from Baseline to Post-Treatment in the Beliefs about Obese People Scale (BAOP) Total Score- Patient | Baseline, Post-Treatment (on average 6 months after beginning treatment)
  8-item self-report scale assessing beliefs about the controllability of obesity.
Change from Baseline to 3-Month Follow-up in the Beliefs about Obese People Scale (BAOP) Total Score- Patient | Baseline, 3-Month Follow-up
  8-item self-report scale assessing beliefs about the controllability of obesity.
Change from Baseline to Post-Treatment in the Attitudes Towards Obese People (ATOP) Total Score- Patient | Baseline, Post-Treatment (on average 6 months after beginning treatment)
  20-item self-report scale assessing perceptions and attitudes about obese people.
Change from Baseline to 3-Month Follow-up in the Attitudes Towards Obese People (ATOP) | Baseline, 3-Month Follow-up
  20-item self-report scale assessing perceptions and attitudes about obese people.
Change from Baseline to Post-Treatment in the Beck Depression Inventory-II Scale (BDI) Total Score- Patient | Baseline, Post-Treatment (on average 6 months after beginning treatment)
  21-item self-report scale assessing severity of current depressive symptoms.
Change from Baseline to 3-Month Follow-up in the Beck Depression Inventory-II (BDI-II) Total Score- Patient | Baseline, 3-Month Follow-up
  21-item self-report scale assessing severity of current depressive symptoms.
Change from Baseline to Post-Treatment in the Beck Anxiety Inventory Scale (BAI) Total Score- Patient | Baseline, Post-Treatment (on average 6 months after beginning treatment)
  21-item self-report scale assessing severity of current anxiety symptoms.
Change from Baseline to 3-Month Follow-up in the Beck Anxiety Inventory Scale (BAI) Total Score- Patient | Baseline, 3-Month Follow-up
  21-item self-report scale assessing severity of current anxiety symptoms.
Change from Baseline to Post-Treatment in the Difficulties in Emotion Regulation Scale (DERS) Total Score- Patient | Baseline, Post-Treatment (on average 6 months after beginning treatment)
  36-item self-report scale assessing four key areas in emotion regulation: 1) awareness and understanding, 2) acceptance of emotions, 3) ability to control impulsive behaviors when having negative emotions, and 4) ability to use emotion regulation strategies.
Change from Baseline to 3-Month Follow-up in the Difficulties in Emotion Regulation Scale (DERS) Total Score- Patient | Baseline, 3-Month Follow-up
  36-item self-report scale assessing four key areas in emotion regulation: 1) awareness and understanding, 2) acceptance of emotions, 3) ability to control impulsive behaviors when having negative emotions, and 4) ability to use emotion regulation strategies.
Change from Baseline to Post-Treatment in the 12-Item Short Form Health Survey (SF-12) Physical Component Summary (PCS)- Patient | Baseline, Post-Treatment (on average 6 months after beginning treatment)
  12-item self-report scale assessing eight different items of functioning over the last month: physical functioning, energy/vitality, bodily pain, social functioning, role limitations due to emotional problems, mental health, and general health.
Change from Baseline to 3-Month Follow-up in the 12-Item Short Form Health Survey (SF-12) Physical Component Summary (PCS)- Patient | Baseline, 3-Month Follow-up
  12-item self-report scale assessing eight different items of functioning over the last month: physical functioning, energy/vitality, bodily pain, social functioning, role limitations due to emotional problems, mental health, and general health.
Change from Baseline to Post-Treatment in the 12-Item Short Form Health Survey (SF-12) Mental Component Summary (MCS)- Patient | Baseline, Post-Treatment (on average 6 months after beginning treatment)
  12-item self-report scale assessing eight different items of functioning over the last month: physical functioning, energy/vitality, bodily pain, social functioning, role limitations due to emotional problems, mental health, and general health.
Change from Baseline to 3-Month Follow-up in the 12-Item Short Form Health Survey (SF-12) Mental Component Summary (MCS)- Patient | Baseline, 3-Month Follow-up
  12-item self-report scale assessing eight different items of functioning over the last month: physical functioning, energy/vitality, bodily pain, social functioning, role limitations due to emotional problems, mental health, and general health.
Change from Baseline to Post-Treatment in the Dyadic Adjustment Scale (DAS) Total Score- Patient | Baseline, Post-Treatment (on average 6 months after beginning treatment)
  32-item self-report scale assessing the quality of the relationship perceived by participants
Change from Baseline to 3-Month Follow-up in the Dyadic Adjustment Scale (DAS) Total Score- Patient | Baseline, 3-Month Follow-up
  32-item self-report scale assessing the quality of the relationship perceived by participants
Change from Baseline to Post-Treatment in the Dyadic Adjustment Scale (DAS) Total Score- Partner | Baseline, Post-Treatment (on average 6 months after beginning treatment)
  32-item self-report scale assessing the quality of the relationship perceived by participants
Change from Baseline to 3-Month Follow-up in the Dyadic Adjustment Scale (DAS) Total Score- Partner | Baseline, 3-Month Follow-up
  32-item self-report scale assessing the quality of the relationship perceived by participants
Change from Baseline to Post-Treatment in the Communication Patterns Questionnaire Short Form (CPQ-SF) Total Score- Patient | Baseline, Post-Treatment (on average 6 months after beginning treatment)
  11-item self-report scale assessing how couple communicates about eating and binge eating disorder.
Change from Baseline to 3-Month Follow-up in the Communication Patterns Questionnaire Short Form (CPQ-SF) Total Score- Patient | Baseline, 3-Month Follow-up
  11-item self-report scale assessing how couple communicates about eating and binge eating disorder.
Change from Baseline to Post-Treatment in the Communication Patterns Questionnaire Short Form (CPQ-SF) Total Score- Partner | Baseline, Post-Treatment (on average 6 months after beginning treatment)
  11-item self-report scale assessing how couple communicates about eating and binge eating disorder.
Change from Baseline to 3-Month Follow-up in the Communication Patterns Questionnaire Short Form (CPQ-SF) Total Score- Partner | Baseline, 3-Month Follow-up
  11-item self-report scale assessing how couple communicates about eating and binge eating disorder.
Change from Baseline to Post-Treatment in the Marital Satisfaction Inventory-Revised (MSI-R) Problem Solving Communication (PSC)- Patient | Baseline, Post-Treatment (on average 6 months after beginning treatment)
  32-item self-report scale assessing communication between partners. The measure has two subscales: Problem Solving Communication (PSC) and Affective Communication (AFC). The 19 true-false items on the PSC reflect three domains: difficulty resolving minor differences, lack of problem solving skills, and inability to discuss sensitive issues. The 13 true-false items on the AFC reflect two dimensions: lack of support/affection and limited disclosure of feelings or lack of understanding.
Change from Baseline to 3-Month Follow-up in the Marital Satisfaction Inventory-Revised (MSI-R) Problem Solving Communication (PSC)- Patient | Baseline, 3-Month Follow-up
  32-item self-report scale assessing communication between partners. The measure has two subscales: Problem Solving Communication (PSC) and Affective Communication (AFC). The 19 true-false items on the PSC reflect three domains: difficulty resolving minor differences, lack of problem solving skills, and inability to discuss sensitive issues. The 13 true-false items on the AFC reflect two dimensions: lack of support/affection and limited disclosure of feelings or lack of understanding.
Change from Baseline to Post-Treatment in the Marital Satisfaction Inventory-Revised (MSI-R) Problem Solving Communication (PSC)- Partner | Baseline, Post-Treatment (on average 6 months after beginning treatment)
  32-item self-report scale assessing communication between partners. The measure has two subscales: Problem Solving Communication (PSC) and Affective Communication (AFC). The 19 true-false items on the PSC reflect three domains: difficulty resolving minor differences, lack of problem solving skills, and inability to discuss sensitive issues. The 13 true-false items on the AFC reflect two dimensions: lack of support/affection and limited disclosure of feelings or lack of understanding.
Change from Baseline to 3-Month Follow-up in the Marital Satisfaction Inventory-Revised (MSI-R) Problem Solving Communication (PSC)- Partner | Baseline, 3-Month Follow-up
  32-item self-report scale assessing communication between partners. The measure has two subscales: Problem Solving Communication (PSC) and Affective Communication (AFC). The 19 true-false items on the PSC reflect three domains: difficulty resolving minor differences, lack of problem solving skills, and inability to discuss sensitive issues. The 13 true-false items on the AFC reflect two dimensions: lack of support/affection and limited disclosure of feelings or lack of understanding.
Change from Baseline to Post-Treatment in the Marital Satisfaction Inventory-Revised (MSI-R) Affective Communication (AFC)- Patient | Baseline, Post-Treatment (on average 6 months after beginning treatment)
  32-item self-report scale assessing communication between partners. The measure has two subscales: Problem Solving Communication (PSC) and Affective Communication (AFC). The 19 true-false items on the PSC reflect three domains: difficulty resolving minor differences, lack of problem solving skills, and inability to discuss sensitive issues. The 13 true-false items on the AFC reflect two dimensions: lack of support/affection and limited disclosure of feelings or lack of understanding.
Change from Baseline to 3-Month Follow-up in the Marital Satisfaction Inventory-Revised (MSI-R) Affective Communication (AFC)- Patient | Baseline, 3-Month Follow-up
  32-item self-report scale assessing communication between partners. The measure has two subscales: Problem Solving Communication (PSC) and Affective Communication (AFC). The 19 true-false items on the PSC reflect three domains: difficulty resolving minor differences, lack of problem solving skills, and inability to discuss sensitive issues. The 13 true-false items on the AFC reflect two dimensions: lack of support/affection and limited disclosure of feelings or lack of understanding.
Change from Baseline to Post-Treatment in the Marital Satisfaction Inventory-Revised (MSI-R) Affective Communication (AFC)- Partner | Baseline, Post-Treatment (on average 6 months after beginning treatment)
  32-item self-report scale assessing communication between partners. The measure has two subscales: Problem Solving Communication (PSC) and Affective Communication (AFC). The 19 true-false items on the PSC reflect three domains: difficulty resolving minor differences, lack of problem solving skills, and inability to discuss sensitive issues. The 13 true-false items on the AFC reflect two dimensions: lack of support/affection and limited disclosure of feelings or lack of understanding.
Change from Baseline to 3-Month Follow-up in the Marital Satisfaction Inventory-Revised (MSI-R) Affective Communication (AFC)- Partner | Baseline, 3-Month Follow-up
  32-item self-report scale assessing communication between partners. The measure has two subscales: Problem Solving Communication (PSC) and Affective Communication (AFC). The 19 true-false items on the PSC reflect three domains: difficulty resolving minor differences, lack of problem solving skills, and inability to discuss sensitive issues. The 13 true-false items on the AFC reflect two dimensions: lack of support/affection and limited disclosure of feelings or lack of understanding.
Change from Baseline to Post-Treatment in the Accommodation and Enabling Scale for Eating Disorders (AESED)- Partner | Baseline, Post-Treatment (on average 6 months after beginning treatment)
  30-item self-report scale assessing accommodating and enabling behaviors of caregivers of people with eating disorders, including subscales for avoidance, modifying routines, reassurance seeking, meal rituals, control of family, and turning a blind eye. Measure edited to be specific to the significant other.
Change from Baseline to 3-Month Follow-up in the Accommodation and Enabling Scale for Eating Disorders (AESED)- Partner | Baseline, 3-Month Follow-up
  30-item self-report scale assessing accommodating and enabling behaviors of caregivers of people with eating disorders, including subscales for avoidance, modifying routines, reassurance seeking, meal rituals, control of family, and turning a blind eye. Measure edited to be specific to the significant other.
Change from Baseline to Post-Treatment in the Beliefs about Obese People Scale (BAOP) Total Score- Partner | Baseline, Post-Treatment (on average 6 months after beginning treatment)
  8-item self-report scale assessing beliefs about the controllability of obesity.
Change from Baseline to 3-Month Follow-up in the Beliefs about Obese People Scale (BAOP) Total Score- Partner | Baseline, 3-Month Follow-up
  8-item self-report scale assessing beliefs about the controllability of obesity.
Change from Baseline to Post-Treatment in the Attitudes Towards Obese People (ATOP) Total Score- Partner | Baseline, Post-treatment (on average 6 months after beginning treatment)
  20-item self-report scale assessing perceptions and attitudes about obese people.
Change from Baseline to 3-Month Follow-up in the Attitudes Towards Obese People (ATOP) Total Score- Partner | Baseline, 3-Month Follow-up
  20-item self-report scale assessing perceptions and attitudes about obese people.
Change from Baseline to Post-Treatment in the Beck Depression Inventory-II Scale (BDI-II) Total Score- Partner | Baseline, Post-Treatment (on average 6 months after beginning treatment)
  21-item self-report scale assessing severity of current depressive symptoms.
Change from Baseline to 3-Month Follow-up in the Beck Depression Inventory-II Scale (BDI-II) Total Score- Partner | Baseline, 3-Month Follow-up
  21-item self-report scale assessing severity of current depressive symptoms.
Change from Baseline to Post-Treatment in the Beck Anxiety Inventory Scale (BAI) Total Score- Partner | Baseline, Post-Treatment (on average 6 months after beginning treatment)
  21-item self-report scale assessing severity of current anxiety symptoms.
Change from Baseline to 3-Month Follow-up in the Beck Anxiety Inventory Scale (BAI) Total Score- Partner | Baseline, 3-Month Follow-up
  21-item self-report scale assessing severity of current anxiety symptoms.
Change from Baseline to Post-Treatment in the Difficulties in Emotion Regulation Scale (DERS) Total Score- Partner | Baseline, Post-Treatment (on average 6 months after beginning treatment)
  36-item self-report scale assessing four key areas in emotion regulation: 1) awareness and understanding, 2) acceptance of emotions, 3) ability to control impulsive behaviors when having negative emotions, and 4) ability to use emotion regulation strategies.
Change from Baseline to 3-Month Follow-up in the Difficulties in Emotion Regulation Scale (DERS) Total Score- Partner | Baseline, 3-Month Follow-up
  36-item self-report scale assessing four key areas in emotion regulation: 1) awareness and understanding, 2) acceptance of emotions, 3) ability to control impulsive behaviors when having negative emotions, and 4) ability to use emotion regulation strategies.

CONTACTS AND LOCATIONS:
Overall Officials: Cristin D Runfola, Ph.D., Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- UNC Center of Excellence for Eating Disorders, Chapel Hill, North Carolina, United States